CLINICAL TRIAL: NCT01488591
Title: Biomarker Research for Personalized Medicine in Blood Cancer Patient
Brief Title: Biomarker Research for Personalized Medicine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Department of Pharmacology and Pharmacogenomics Research Center, Inje University
Other Study IDs: 09-029
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study :

1. Through the study of genes of protein, transporter, translator and epigenome investigating the effect of anti-cancer treatment or the key factor of the MDR (Multidrug resistance) on the blood cancer patients who are under the anti-cancer sork treatment
2. Giving a service of anticancer medicine therapeutic drug monitoring (TDM) and genotyping

ELIGIBILITY:
Inclusion Criteria:

* Korean
* Clinical diagnosis of Hematologic neoplasms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University, Busan, South Korea